CLINICAL TRIAL: NCT02637752
Title: Efficacy of Nutrition and Physical Activity Counselling for Pre-adolescent Children in a Dental Setting: A Randomized Clinical Trial
Brief Title: Nutrition and Physical Activity Counselling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Amir Azarpazhooh, Dr., University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMAZ 515
Record Dates: First submitted 2015-12-14; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Childhood Obesity
Keywords: Pediatric Obesity; Body Mass Index; Dentistry
MeSH Terms: conditions — Pediatric Obesity | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Active Comparator): Intervention: Lifestyle counseling or nutrition/physical counselling
  Interventions: Behavioral: Lifestyle counseling or nutrition/physical counselling
- No Intervention (No Intervention): To ensure that both groups benefited equally from the study, the control group received the counselling and the handouts at the end of the study.

INTERVENTIONS:
Behavioral: Lifestyle counseling or nutrition/physical counselling — A brief (5-10 minute) counseling session for caregivers of the intervention group aimed to encourage an increase in the child's physical activity and decrease sugar-sweetened beverage consumption and screen time. Additionally, the caregivers of the intervention group were provided with the following handouts: five steps to a healthy body weight for teens; beverages; physical activity tips for children 5-11 years; Canadian physical activity guidelines for children 5-11; and Canadian sedentary behavior guidelines for children 5-11.
  Arms: Lifestyle counseling

SUMMARY:
Background: Childhood obesity imposes a great burden on the healthcare system. Given the increased frequency of dental compared to medical visits during childhood, dentists may be in an ideal position to recognize patients at risk of developing obesity. This randomized clinical trial explored the efficacy of a brief nutrition and physical activity counseling for healthy weight 6 to11 year-old children in a university-based pediatric dental clinic.

Methods: 168 children, 6-11 year old, were allocated to test and control groups and their Body Mass index (BMI) were recorded. Their parents/caregivers completed a questionnaire regarding their child's nutrition, physical activity and screen time. The parents/caregivers of the test group then received a brief counseling session that encouraged an increase in children's physical activity, and a decrease in sugar-sweetened beverages and screen time. Data, collected at baseline and follow-up session (within 6-12 months) were analyzed using general linear regression, adjusting for age, gender, socio-demographic characteristics, education, labour force, income and awareness of school nutrition policy (P≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* healthy
* 6 to 11 years old

Exclusion Criteria:

* Younger or older children
* those with systemic diseases (such as diabetes, cardiac problems, dyslipidemia, elevated cholesterol, obstructive sleep apnea, stroke, fatty liver disease, osteoarthritis, orthopedic problems and any forms of cancer)
* Children and their accompanying parents or caregivers (hereafter, caregivers) unable to communicate in English
* if caregivers were unreachable after three attempts by phone

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 6-12 months from the baseline

SECONDARY OUTCOMES:
physical activity (hrs/day) | 6-12 months
screen time (hrs/day) | 6-12 months
number of sugar-sweetened beverages consumed per day | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Amir Azarpazhooh, DDS MSc PhD, Principal Investigator — Assistant Professor

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Azarpazhooh A, Sekhavat A, Sigal MJ. Validity of a simplified screening instrument for assessing overweight children in a dental setting: a cross sectional study. BMC Pediatr. 2017 Feb 17;17(1):56. doi: 10.1186/s12887-017-0808-x. PMID 28212686